CLINICAL TRIAL: NCT04765995
Title: A Study to Investigate the Pharmacokinetics, Safety, Tolerability and Immunogenicity of HZBio1 in Healthy Chinese Volunteers
Brief Title: Study of Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of of HZBio1 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Grand Biologic Pharmaceutical, Inc. (Industry)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YDHY（HZBio1）-001（I）
Record Dates: First submitted 2021-01-12; First posted 2021-02-23 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- HZBio1 0.96mg/kg (Experimental): Participants will receive intramuscularly 0.96 milligram per kilogram (mg/kg) of HZBio1.
  Interventions: Drug: HZBio1 0.96mg / kg; Drug: Placebo
- HZBio1 3mg/kg (Experimental): Participants will receive intramuscularly 3 milligram per kilogram (mg/kg) of HZBio1.
  Interventions: Drug: HZBio1 3mg / kg; Drug: Placebo
- HZBio1 6mg/kg (Experimental): Participants will receive intramuscularly 6 milligram per kilogram (mg/kg) of HZBio1.
  Interventions: Drug: HZBio1 6mg / kg; Drug: Placebo
- HZBio1 9mg/kg (Experimental): Participants will receive intramuscularly 9milligram per kilogram (mg/kg) of HZBio1.
  Interventions: Drug: HZBio1 9mg / kg; Drug: Placebo
- HZBio1 12mg/kg (Experimental): Participants will receive intramuscularly 12 milligram per kilogram (mg/kg) of HZBio1.
  Interventions: Drug: HZBio1 12mg / kg; Drug: Placebo

INTERVENTIONS:
Drug: HZBio1 0.96mg / kg — HZBio1 will be administered intramuscularly in single ascending doses with starting of 0.96 mg/kg and subsequent doses of 3.0 mg/kg, 6.0 mg/kg ,9.0 mg/kg,and 12mg/kg, respectively.
  Arms: HZBio1 0.96mg/kg
Drug: HZBio1 3mg / kg — HZBio1 will be administered intramuscularly in single ascending doses with starting of 0.96 mg/kg and subsequent doses of 3.0 mg/kg, 6.0 mg/kg ,9.0 mg/kg,and 12mg/kg, respectively.
  Arms: HZBio1 3mg/kg
Drug: HZBio1 6mg / kg — HZBio1 will be administered intramuscularly in single ascending doses with starting of 0.96 mg/kg and subsequent doses of 3.0 mg/kg, 6.0 mg/kg ,9.0 mg/kg,and 12mg/kg, respectively.
  Arms: HZBio1 6mg/kg
Drug: HZBio1 9mg / kg — HZBio1 will be administered intramuscularly in single ascending doses with starting of 0.96 mg/kg and subsequent doses of 3.0 mg/kg, 6.0 mg/kg ,9.0 mg/kg,and 12mg/kg, respectively.
  Arms: HZBio1 9mg/kg
Drug: HZBio1 12mg / kg — HZBio1 will be administered intramuscularly in single ascending doses with starting of 0.96 mg/kg and subsequent doses of 3.0 mg/kg, 6.0 mg/kg ,9.0 mg/kg,and 12mg/kg, respectively.
  Arms: HZBio1 12mg/kg
Drug: Placebo — Matching placebo will be administered intramuscularly.

SUMMARY:
This randomized study will evaluate the safety, tolerability ,pharmacokinetics, pharmacodynamics and Immunogenicity of single ascending intramuscularly administered doses of HZBio1 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed and signed informed consent form;
2. Healthy subjects, male and female;
3. At the time of signing the informed consent, they were over 18-45 years old (including 18 and 45 years old) and weighed more than 50 kg,

   Body mass index ranged from 19 to 26 (including 19 and 26) [body mass index (BMI) = body weight (kg) / height 2 (M2)];
4. The results of serum pregnancy test in women of childbearing age were negative;
5. The subjects agreed to use effective contraception or abstinence during the study period and within 6 months after the end of the study;
6. Be able to understand and comply with the clinical protocol requirements, and it is expected to complete the whole trial process.

Exclusion Criteria:

1. History of hypertension or abnormal blood pressure at screening / baseline (SBP > 140 mmHg and / or DBP > 90 mmHg confirmed twice a day)
2. According to the researcher's judgment (clinical urine routine examination, proteinuria 2 + and above), proteinuria or proteinuria history with clinical significance.
3. Any previous VEGF and VEGFR antibody or protein therapy within one year.
4. No biological products or live virus vaccine shall be used for treatment for 3 months before the first administration of the study drug, or any monoclonal antibody shall be used for 12 months.
5. History or evidence of hereditary bleeding, coagulopathy, or thrombosis.
6. History of gastrointestinal perforation or fistula.
7. Severe, unhealed wounds, active ulcers, or untreated fractures, or were randomly assigned or expected to require major surgery during the course of the study or within 2 months after the last administration of the study drug.
8. RX or OTC drugs or nutritional supplements were used within 5 half lives before the first administration of the study drug or within 2 weeks (depending on the longer period). Herbal supplements need to be discontinued 28 days before the first administration of the study drug.
9. HBsAg, HCV antibody, HIV antibody and syphilis were positive
10. Known allergy to bevacizumab or any excipient
11. Known allergic diseases or allergic constitution
12. There was a history of unpaid blood donation within 3 months before taking the study drug for the first time
13. Use any other study drug for treatment or participate in other clinical trials within 3 months before screening
14. There was a history of alcohol or drug abuse within 12 months before screening; subjects were not able to control within 72 hours before and throughout the study
15. History of mental illness
16. During the study, the partner was expected to be pregnant.
17. During the study period, it did not conform to the clinical study protocol.
18. Other conditions not suitable for this study were considered by the researchers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | 36 days
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Tmax of HZBio1 | 36 days
  Time to peak (Tmax)
Cmax of HZBio1 | 36 days
  peak concentration (Cmax)
Кel of HZBio1 | 36 days
  Кel of HZBio1 (elimination constant)
Т1/2 of HZBio1 | 36 days
  Т1/2 of HZBio1 (half-life)
AUC0-t of HZBio1 | 36 days
  AUC0-t of HZBio1 (the area under the Concentration vs. Time curve from 0 to t post-infusion)
serum uric acid level | 36 days
  The decrease of serum uric acid level after administration will be analyzed.
Number of Participants Positive for Nab（Neutralizing Antibody） | 36 days
  The changes of neutralizing antibody were observed before and after treatment.
Number of anti peg antibody | 36 days
  The changes of anti peg antibody were observed before and after treatment.
Number of anti PHC antibody | 36 days
  The changes of anti PHC antibody were observed before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhong Liu, Principal Investigator — Peking Union Medical College Hospital; Xin Zheng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China